CLINICAL TRIAL: NCT01413074
Title: A Prospective, Randomized, Multicenter, Open-Label, Interventional Study Comparing Survival in Subjects Receiving Peritoneal Dialysis vs Hemodialysis in China
Brief Title: Survival on Peritoneal Dialysis (PD) Versus Hemodialysis (HD) in China
Status: Terminated | Phase: Phase 4 | Type: Interventional
Sponsor: Baxter Healthcare Corporation (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CHN-RENAL-CTPIV-2010-106
Record Dates: First submitted 2011-06-16; First posted 2011-08-10 (Estimated); Last update posted 2016-05-19 (Estimated); Status verified 2016-05

CONDITIONS: End Stage Renal Disease
Keywords: End Stage Renal Disease; ESRD; Peritoneal Dialysis; PD; Hemodialysis; HD
MeSH Terms: conditions — Kidney Failure, Chronic

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- ESRD patients receiving HD treatment (Active Comparator): no investigational drug involved. Only oberseve therapy treatment
  Interventions: Other: Hemodialysis treatment
- ESRD patients receiving PD treatment (Experimental): no investigational drug involved. Only oberseve therapy treatment
  Interventions: Other: Peritoneal Dialysis treatment

INTERVENTIONS:
Other: Peritoneal Dialysis treatment — PD treatment
  Arms: ESRD patients receiving PD treatment
Other: Hemodialysis treatment — HD treatment
  Arms: ESRD patients receiving HD treatment

SUMMARY:
Primary Objective: The primary objective is to prospectively assess and compare survival in subjects with End Stage Renal Disease (ESRD) randomized to Peritoneal Dialysis (PD) or Hemodialysis (HD) treatment.

Secondary Objectives: The secondary objectives are to prospectively assess and compare the following parameters in subjects receiving PD or HD treatment:

* Technique failure
* Cause of death
* Comorbidity status at baseline and changes throughout the study
* Change in residual renal function (RRF)
* Dialysis adequacy (i.e., Kt/Vurea)
* Change in blood pressure, hemoglobin, and S-phosphate
* Change in nutritional status
* Occurrence of bacterial and other infections
* Hospitalization, including number, duration, and underlying reason(s)
* Systemic inflammation as assessed by high-sensitivity C reactive protein (hs-CRP)
* Quality of life (QOL)

Safety Objectives: To compare the nature and frequency of adverse events (AEs) and serious adverse events (SAEs), including abnormal laboratory test findings with clinical significance, in subjects receiving PD or HD treatment.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects of either sex, aged 18 years or older at time of randomization.
2. Subjects diagnosed with ESRD (glomerular filtration rate [GFR] ≤ 15 mL/min/m2 body surface area [BSA]) and predicted by the investigator to need dialysis therapy within 10 weeks after the pre-screening period.
3. Subjects who, as judged by the investigator, are able to comprehend the pre-defined, standardized, modality education program and have undertaken this education during the screening period.
4. Subjects, or their legal representative, who, as judged by the investigator, are capable of being trained for home-based PD.
5. Subjects, or their legal representative, who are able to understand and voluntarily sign an ICF.
6. Subjects who are able to adhere to the study visit schedule and other protocol requirements.
7. Subjects who are able to regularly visit a HD center for HD therapy (≥ 3 times per week).
8. Subjects who, as judged by the investigator, are expected to remain on dialysis for at least 48 weeks.
9. Subjects who have normal liver function, as judged by the investigator.
10. Female subjects of childbearing potential who have a negative serum or urine pregnancy test at screening. Sexually active women of childbearing potential must agree to use adequate contraceptive methods, as judged by the investigator, while in the study.

Exclusion Criteria:

1. Subjects who are HIV positive.
2. Subjects who have already received a permanent PD catheter or HD access that is intended for permanent use before receiving modality education or have already received permanent dialysis. Subjects are not excluded if an access is present within 4 weeks before screening for back-up purposes or for acute treatment of life-threatening uremic symptoms, electrolyte abnormalities, or fluid overload.
3. Subjects who have a serious, uncontrolled medical disorder or active infection, which, as judged by the investigator, would jeopardize their ability to receive the prescribed dialysis treatment.
4. Subjects who have dementia or a mental status that would significantly affect the subject's understanding of the Informed Consent Form (ICF).
5. Subjects who are pregnant, intend to become pregnant during the study period, or are breast-feeding.
6. Subjects with a history of drug (defined as illicit drug use) or alcohol (defined as regular or daily consumption of more than 4 alcoholic drinks per day) abuse in the 2 years before screening.
7. Subjects who have previously received renal transplantation and are still being prescribed immunosuppressive therapy.
8. Subjects who are currently using or have used an investigational product within five half-lives of the physiological action or 30 days, whichever is longer, before screening.
9. Subjects who are unwilling or expected to be unable to fully comply with the visits and assessments required by the protocol.
10. Subjects who have previously been randomized in this study.
11. Subjects who are not eligible for either PD or HD, as judged by the investigator, due to:

    PD: documented extensive intra-peritoneal adhesions or other condition contraindicated for PD.

    HD: severe cardiac instability or other condition contraindicated for HD.
12. Subjects who have a serious or acute condition that, as judged by the investigator, would preclude participation in the study.
13. Subjects who have a malignancy requiring chemotherapy or radiation therapy.
14. Subjects undergoing temporary dialysis treatment between the screening visit and Day 1 that is expected to exceed 6 weeks in duration.
15. Subjects who have a life expectancy of less than 48 weeks.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 416 (Actual)
Dates: Start 2011-06; Primary Completion 2013-12 (Actual); Study Completion 2013-12 (Actual)

PRIMARY OUTCOMES:
Assess and compare survival or all cause mortality in subjects undergoing PD or HD treatment | 2-5 yrs.

SECONDARY OUTCOMES:
Assess and compare technique failure | 2-5 yrs.
  Technique failure is defined as a change of dialysis modality (PD to HD, or HD to PD) or death. However, a temporary transfer, defined as ≤ 6 weeks duration and ≤ 2 occasions per any 52-week period, will not be considered technique failure. The use of both modalities within a 7-day period for more than 4 consecutive weeks will be considered technique failure. Technique failure will be monitored in two ways: modality failure including deaths and technique failure not including deaths.
Residual Renal Function (RRF) | 2-5 yrs
  RRF will be estimated if the subject's urine volume is ≥ 100 mL/24 h. RRF will be assessed by calculating GFR from a 24-h urine urea and creatinine collection and normalized to 1.73 m2 Body Surface Area. RRF will be measured at screening, visit 1 and every 12 weeks after visit 1 till the end of the study. Subjects who have a permanent modality transfer will be followed up for RRF (with the frequency of assessment determined by the modality they are switched to) until the end of the study, transplantation, stopping dialysis, lost to follow-up, or death.
Dialysis Adequacy | 2-5 yrs.
  In subjects receiving PD, dialysis adequacy (Kt/Vurea) will be assessed at 4 weeks (visit 2), 12 weeks (visit 4) and then every 12 weeks (±14 days) until the end of the study (±14 days). Kt/Vurea target for PD patients is ≥ 1.7 per week. Kt/Vurea target for HD patients is ≥ 1.2 per dialysis session. Subjects who have a permanent modality transfer will be followed up for Kt/Vurea (with the frequency of assessment determined by the modality they are switched to) until the end of the study, transplantation, stopping dialysis, lost to follow-up, or death.
Co-morbidity Assessment | 2-5 yrs.
  The Charlson Comorbidity Index contains 19 categories of comorbidity which are primarily defined using ICD-9-CM diagnoses codes, as well as a few procedure codes. The overall comorbidity score reflects the cumulative increased likelihood of one-year survival; the higher the score, the more severe the burden of comorbidity. Every diagnosis and procedure code is analyzed to see if it falls within one of the 16 comorbid conditions. In this study, the comorbidity assessment will be measured at visit 1, every 24 weeks (±14 days) after visit 1 to visit 23, and at the end-of-study visit.
Occurrence of Bacterial and Other Infections Infection rates | 2-5 yrs.
  Occurrence of bacterial and other infections infection rates, especially regarding exit sites and peritoneal, will be monitored for HD and PD patients.
Hospitalization | 2-5 yrs.
  Hospitalization rates and duration for each underlying reason will be monitored for HD and PD patients.
Transplantation Rate | 2-5 yrs.
  Kidney transplantation is the best outcome that a patient can expect. By default, a patient will be discontinued from the study after transplantation. Imbalance of the transplantation rate between HD and PD will be assessed. However, all patients will be followed to the end of the study to assess the primary endpoint which is all-cause mortality.
Cause of Death | 2-5 yrs.
  Cause of deaths due to acute myocardial infarction (AMI), congestive heart failure (CHF), infection (except peritonitis), peritonitis, malnutrition, stroke, cardiovascular and non-cardiovascular causes, etc., will be monitored for HD and PD patients
Change in Erythropoiesis-stimulating agent (ESA) | 2-5 yrs.
  Dose changes in ESA dose will affect patient's status for anemia control, and will be monitored for HD and PD patients.
Change in blood pressure, hemoglobin, and S-phosphate | 2-5 yrs.
  Blood pressure, hemoglobin, and S-phosphate will be monitored for HD and PD patients.
Subjective Global Assessment for Nutritional Status | 2-5 yrs.
  Subjective Global Assessment (SGA) is a technique to assess a patient's nutritional status. The SGA will be measured by one dedicated, trained physician per site at visit 1, every 24 weeks (±14 days) from visit 1 to visit 23, and at the end-of-study visit.
Systemic inflammation as assessed by hs-CRP | 2-5 yrs.
  Scores of systemic inflammation will be assessed using high-sensitivity C reactive protein (hs-CRP). Hs-CRP will be assessed at visits 1, 4-23, and at the end-of-study visit.
Quality of Life Quality of life (QOL) | 2-5 yrs.
  Quality of Life Quality of life (QOL) will be assessed using the EQ-5D-3L (European Quality of Life - 5 Dimensions - 3L translation), the KDQoL-SF (Kidney Disease Quality of Life Short Form) questionnaires, and the Karnofsky Index. QOL will be assessed at visit 1, every 24 weeks (±14 days) from visit 1 to visit 23, and at the end-of-study visit.

CONTACTS AND LOCATIONS:
Overall Officials: Quian Jia-Qi, Prof., Principal Investigator — Shanghai Jiao Tong University School of Medicine; Yu Xue-qing, Prof., Principal Investigator — First Affiliated Hospital, Sun Yat-Sen University
Locations (7):
- China (7):
  - The First Affiliated Hospital , Sun Yet-Sen University, Guangzhou, Guangdong
  - Shanghai Changzheng Hospital, Shanghai, Shanghai Municipality
  - Ruijin Hospital,Shanghai Jiaotong University , School of Medicine, Shanghai, Shanghai Municipality
  - Huashan Hospital ,Fudan University, Shanghai, Shanghai Municipality
  - Renji Hospital , Shanghai Jiaotong University , School of Medicine, Shanghai, Shanghai Municipality
  - The First Affiliated Hospital , Zhejiang University, School of Medicine, Hangzhou, Zhejiang
  - Hangzhou Hospital of Tranditional Chinese Medicine, Hangzhou, Zhejiang

REFERENCES:
- [Derived] Ethier I, Hayat A, Pei J, Hawley CM, Johnson DW, Francis RS, Wong G, Craig JC, Viecelli AK, Htay H, Ng S, Leibowitz S, Cho Y. Peritoneal dialysis versus haemodialysis for people commencing dialysis. Cochrane Database Syst Rev. 2024 Jun 20;6(6):CD013800. doi: 10.1002/14651858.CD013800.pub2. PMID 38899545
- [Derived] Quinn RR, Lam NN. Home Dialysis in North America: The Current State. Clin J Am Soc Nephrol. 2023 Oct 1;18(10):1351-1358. doi: 10.2215/CJN.0000000000000273. Epub 2023 Jul 31. PMID 37523194